CLINICAL TRIAL: NCT04595344
Title: Effects of Listening to Binaural Beats on Anxiety Levels and Pain Scores in Male Patients Undergoing Cystoscopy and Ureteral Stent Removal: A Randomized Placebo-controlled Trial
Brief Title: Effects of Listening to Binaural Beats on Anxiety and Pain Scores in Males Undergoing Cystoscopy and Stent Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mahmut Taha Olcucu, Asst. Prof., Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16/15
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Anxiety; Cystoscopy; Pain
Keywords: Anxiety; Binaural beats; Cystoscopy; Pain; Ureteral Stent Removal
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Diagnostic cystoscopy , Binaural beat group (Active Comparator): patients listened to binaural beats
  Interventions: Other: Listening to Pure Binaural Beats
- Diagnostic cystoscopy, Classical music group (Active Comparator): patients listened to classical music
  Interventions: Other: Listening to classical music
- Diagnostic cystoscopy , Placebo group (Placebo Comparator): patients no audio only headphones
  Interventions: Other: No audio only headphone
- Ureteral stent removal, Binaural beat group (Active Comparator): patients listened to binaural beats
  Interventions: Other: Listening to Pure Binaural Beats
- Ureteral stent removal ,Classical music group (Active Comparator): patients listened to classical music
  Interventions: Other: Listening to classical music
- Ureteral stent removal, Placebo group (Placebo Comparator): patients no audio only headphones
  Interventions: Other: No audio only headphone

INTERVENTIONS:
Other: Listening to Pure Binaural Beats — The patients in DCG ((binaural beat group) ) and USRG (binaural beat group) listened to binaural beats.The binaural beats were produced using a software program (Audacity®, version win. 2.3.2, 2019 Audacity Team) at frequency of 10 Hz (a tone of 200 Hz in the right ear and a tone of 210 Hz in the left ear). The binaural beats that the patients in DCG-1 and USRG-1 listened to were "pure" frequencies, with no background music or waves.
  Arms: Diagnostic cystoscopy , Binaural beat group; Ureteral stent removal, Binaural beat group
Other: Listening to classical music — The patients in DCG (classical music group) and USRG (classical music group) listened to classical music.The classical music that those in DCG-2 and USRG-2 listened to was Mozart's 40th Symphony.
  Arms: Diagnostic cystoscopy, Classical music group; Ureteral stent removal ,Classical music group
Other: No audio only headphone — The patients in DCG (placebo group) and USRG (placebo group) sat in a quiet room with headphones on but no audio playing
  Arms: Diagnostic cystoscopy , Placebo group; Ureteral stent removal, Placebo group

SUMMARY:
This study aimed to investigate the effects of pure binaural beats on anxiety levels and pain scores using the State-Trait Anxiety Inventory (STAI) questionnaire and Visual Analog Scale (VAS) in male patients undergoing DC and USR procedures under local anesthesia.

DETAILED DESCRIPTION:
Diagnostic cystoscopy (DC) and ureteral stent removal (USR) are two common simple procedures in urology practice. DC is generally performed to investigate the etiology of hematuria, recurrent urinary tract infections, lower urinary tract symptoms, and suspected bladder tumor cases.Ureteral stent removal is usually carried out after the placed urethral stent for the treatment of urolithiasis and urethral stricture. In many urology clinics, both procedures are generally performed under local anesthesia. To reduce pain, it is recommended that DC should be performed using a flexible cystoscope. In many urology clinics, USR is performed using a rigid cystoscope in both sexes, as a rigid cystoscope is easier to manipulate during stent removal compared with a flexible cystoscope. Although performed under local anesthesia, both procedures are invasive and can cause increased anxiety levels and pain perception.Anxiety is commonly associated with an increased perception of pain.Therefore, patients who have high anxiety levels experience longer pain and require more analgesics.

Binaural beats have been recommended to reduce anxiety levels and the perception of pain in many treatment modalities.hey were discovered by Dove in 1841 and described in detail by Oster in 1973. Binaural beats are resulted from exposing each ear to two sounds which have steady intensities with different frequencies. A single tone with a midway frequency between the carrier tones is perceived. This frequency also waxes and wanes in amplitudes at a rate equal to the difference between the carrier tones It has been suggested that the human brain alters its dominant wave frequency toward that of the frequency of external stimuli to synchronize neural activity with stimuli from binaural beats.

METHOD

Ethics statement and participant selection

The study was approved by the institutional review board (Approval number and date: 16/15 - 04/07/2019 ). Male patients aged ≥ 18 y with negative urine culture, at least formal schooling (1-8 y of education) who had undergone local DC for various reasons (e.g., hematuria, carcinoma suspicion, follow-up for bladder cancer, and screening of the urethra or prostate) or unilateral USR were included in the study. Informed consent was provided by all the patients who accepted to participate in the study.

The exclusion criteria were patients who had a hearing or vision problems, neurological deficits, mental retardation, a history of chronic pelvic pain syndrome, history of previous DC or USR procedures, antidepressant use, or analgesia use 24 h before the procedure. Patients who underwent a bilateral USR procedure (for USR patients), required additional manipulations of the lower urinary tract (e.g., urethral dilation or biopsies), declined to participate, failed to complete the questionnaires, or could not tolerate the intervention were also excluded from the study.

Randomization, sample size, procedures, interventions, measurement of anxiety levels and pain scores

This was a prospective randomized, non-blinded and placebo-controlled study. After initial exclusions, patients were allocated to the study using the block randomization method. Two main groups were created according to the procedure applied: a DC group (DCG) and a USR group (USRG). The patients in the DCG were divided into three subgroups, according to the intervention applied: DCG-1, patients listened to binaural beats; DCG-2, patients listened to classical music; and DCG-3, patients wore headphones but were not exposed to audio (control group). The USRG was also divided into three subgroups, according to the intervention applied: USRG-1 patients listened to binaural beats; USRG-2 patients listened to classical music; and USRG-3 patients wore headphones but were not exposed to audio (control group). A power analysis indicated a minimum of 62 patients were required in each DCG to have power (1-β) of 0.90 at an alpha value of 0.05, with an effect size of 0.265. A minimum of 41 patients was required in each USRG to have power (1-β) of 0.90 at an alpha value of 0.05 with an effect size of 0.326. The sample sizes of the groups were calculated using the G-power 3.1 (Kiel, Germany).

The STAI is a questionnaire used for measuring anxiety.20 The STAI is often employed to determine an individual's emotional status before surgical interventions. It consists of 20 questions, and STAI scores range from 20 to 80. Higher STAI scores indicate increased anxiety levels. In this study, we used the Turkish validation of the STAI questionnaire to evaluate the patients' anxiety scores.21 Before the DC and USR procedures, the patients who accepted to participate in the study were asked to complete the STAI questionnaire and a nurse recorded the score of each patient (initial STAI: STAI-I). All the patients then put on headphones. For 10 min before the interventions, the patients in DCG-1 and USRG-1 listened to binaural beats, those in DCG-2 and USRG-2 listened to classical music and those in DCG-3 and USRG-3 sat in a quiet room with headphones on but no audio playing. The binaural beats were produced using a software program (Audacity®, version win. 2.3.2, 2019 Audacity Team) at frequency of 10 Hz (a tone of 200 Hz in the right ear and a tone of 210 Hz in the left ear). The binaural beats that the patients in DCG-1 and USRG-1 listened to were "pure" frequencies, with no background music or waves. The classical music that those in DCG-2 and USRG-2 listened to was Mozart's 40th Symphony. The audio headphones used in the DCGs and USRGs were wireless stereo headphones (Sony WH-CH510; Sony Corporation, U.S.). The patients who could not tolerate the interventions were also recorded. After the interventions, the STAI scores of the patients were measured again and recorded. (Terminal STAI: STAI-T). Delta anxiety score is recorded as STAI-I score minus STAI-T score (delta STAI: STAI-D).

The genital area was disinfected with povidone-iodine, and 10 ml of 2% lidocaine jelly was instilled intraurethrally and the penis was clamped approximately 5 min for local anesthesia before the procedures. We used a 17 F video flexible cystoscope for DCG procedure (Hawk GmbH, China) and 17 F rigid cystoscope (Stema GmbH, Germany) with 30 ͦ telescope (Karl Storz GmbH, Germany) for USR procedure. Semi-rigid forceps were used when performing USR. During the DC and USR procedures, the same interventions before the procedures were applied to the patients again. The VAS is a common tool in which patients score their pain level on a scale between 0 and 10.22 In this study, we also used the VAS to evaluate the patients' pain scores. After the procedures, the duration of the procedures and VAS scores 20 of the patients were also recorded. The duration of each procedure was calculated as the time between the entry and exit of the cystoscopy device into the urethral meatus.

Statistical Analysis

The Statistical analysis was made using IBM SPSS Statistics for Windows, Version 25.0 (IBM Corp., Armonk, NY). The assumptions of normality were evaluated by the Shapiro-Wilk test. To determine differences between groups, One-way ANOVA test was used for parametric variables and Kruskal Wallis test was used for non-parametric variables. Bonferroni-Dunn test was used as a post-hoc test for significant cases. Pearson chi-square test and Fisher's exact test were used to compare the categorical variables between the groups while Bonferroni-Dunn test was also used as a post-hoc test for significant cases. A p value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* negative urine culture
* at least formal schooling (1-8 y of education)

Exclusion Criteria:

* hearing or vision problems
* neurological deficits
* mental retardation
* history of chronic pelvic pain syndrome
* history of previous DC or USR procedures
* antidepressant use or analgesia use 24 h before the procedure
* decline to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 352 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Binaural beats and anxiety levels | 10 minutes
  Effects of listening to binaural beats on axiety levels before diagnostic cystoscopy and ureteral stent removal procedures. STAI was used to assess the anxiety levels of the patients. STAI scores range from 20 to 80. Higher STAI scores indicate increased anxiety levels
Binaural beats and pain scores | 8 minute
  Effects of listening to binaural beats on pain scores during diagnostic cystoscopy and ureteral stent removal procedures. VAS vas used to assess the pain scores of patients. The VAS is a common tool in which patients score their pain level on a scale between 0 (no pain) and 10 ( worst pain possible).

SECONDARY OUTCOMES:
Classical Music and anxiety levels. | 10 minutes
  Effects of listening to classical music on axiety levels before diagnostic cystoscopy and ureteral stent removal procedures. STAI was used to assess the anxiety levels of the patients.STAI scores range from 20 to 80. Higher STAI scores indicate increased anxiety levels
Classical music and pain scores | 8 minutes
  Effects of listening to classical music on pain scores during diagnostic cystoscopy and ureteral stent removal procedures. VAS vas used to assess the pain scores of patients.he VAS is a common tool in which patients score their pain level on a scale between 0 (no pain) and 10 ( worst pain possible).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Taha MO Ölçücü, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)